CLINICAL TRIAL: NCT04605757
Title: Pulmonary Involvement of Novel SARS-COV-2 Infection (COVID-19): Long-term Impact and Predictors of Possible Lasting Damage: Follow the Covid Study
Brief Title: Long-term Evolution of Pulmonary Involvement of Novel SARS-COV-2 Infection (COVID-19): Follow the Covid Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Stefano Nava, Professor of Respiratory Medicine/ Alma Mater Studiorum University of Bologna (IT)- Director of Respiratory and Critical Care Unit/ S.Orsola-Malpighi University Hospital, Bologna (IT), IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: 714/2020/Oss/AOUBo
Record Dates: First submitted 2020-10-11; First posted 2020-10-28 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: SARS-COV-2 Pneumonia
Keywords: SARS-COV-2
MeSH Terms: interventions — Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute respiratory failure due to SARS-COV-2: Patients admitted to hospital with acute respiratory failure due to SARS-COV-2 infection causing pneumonia
  Interventions: Other: Clinical, functional and radiological lung involvement evolution

INTERVENTIONS:
Other: Clinical, functional and radiological lung involvement evolution — Observational / Clinical, functional and radiological long term evolution of SARS-COV-2 lung involvement

SUMMARY:
In December 2019 the first case of human infection by a new coronavirus was identified, currently called SARS-COV-2 (Severe Acute Respiratory Syndrome - Coronavirus - 2), characterized by high contagiousness and the possibility of causing a severe acute respiratory distress syndrome from which its acronym derives and which caused the state of a global pandemic in a few months. The most frequent clinical manifestation of COVID-19 is pneumonia, which in about 20% of cases results in acute respiratory failure. Very few studies have so far addressed the problem of clinical and functional recovery in these patients, most of them just before or after discharge and none specifically focused on patients admitted for ARF. Indeed most of these investigations were limited to a specific field such as symptoms, pulmonary function and radiological changes. There are no guidelines for the follow-up of COVID-19 patients, despite the British Thoracic Society (BTS) has published a guidance for scheduling post-hospitalization assessments.

Aim of this study is to describe the long term (6 to 12 months) evolution of lung involvement in patients discharged after an episode of ARF due to COVID-19, identifying possible factor associated to lasting clinical, functional or radiological abnormalities collecting data from hospital stay, 1-month after hospital discharge, 3-months after hospital discharge and 6-to-12-months after hospital discharge.

DETAILED DESCRIPTION:
Coronaviruses are a family of viruses with marked tropism for the respiratory system, being able to cause heterogeneous pathological states in humans ranging from the common cold to more serious diseases such as Respiratory Syndrome severe acute respiratory syndrome (SARS). In December 2019 in Wuhan in China, the first case of human infection by a new coronavirus was identified, currently called SARS-COV-2 (Severe Acute Respiratory Syndrome - Coronavirus - 2), characterized by high contagiousness and the possibility of causing a severe acute respiratory distress syndrome from which its acronym derives and which caused the state of a global pandemic in a few months. The disease caused by the SARS-COV-2 virus is called COVID 19.

The most frequent clinical manifestation of COVID-19 is pneumonia, which in about 20% of cases results in acute respiratory failure requiring oxygen therapy or ventilatory support. sometimes resulting in a picture similar to that caused by acute respiratory distress syndrome (ARDS), found in 60-70% of patients admitted to intensive care. The pathogenesis of classical ARDS involves three phases of the disease: an exudative, a proliferative and a fibrotic phase, which occurs when the removal of alveolar collagen fails and leads to progressive pulmonary fibrosis. It is not known whether the long-term evolution of the COVID 19 disease could result in the establishment of a fibrotic phase similar to that predicted by the pathogenesis of classical ARDS, which would lead to a chronic ventilatory deficit similar to that of pulmonary interstitial diseases, with serious impact on quality of life and mortality.

However, it is not well-known whether SARS-COV-2 pneumonia causes restitutio ad integrum or whether it can induce persistent parenchymal alterations and lung function abnormalities.

Very few studies have so far addressed the problem of clinical and functional recovery in these patients, most of them just before or after discharge and none specifically focused on patients admitted for ARF. Indeed most of these investigations were limited to a specific field such as symptoms, pulmonary function and radiological changes.There are no guidelines for the follow-up of COVID-19 patients, despite the British Thoracic Society (BTS) has published a guidance for scheduling post-hospitalization assessments.

Aim of this study, spontaneous,observational, both prospectic and retrospective, is to describe the long term (6 to 12 months) evolution of lung involvement in patients discharged after an episode of ARF due to COVID-19, identifying possible factor associated to lasting clinical, functional or radiological abnormalities.

Investigators will collect clinical, functional and radiological parameters during:

* the hospital stay due to COVID-19 (H);
* the 1-month after hospital discharge followup visit (V1);
* the 3-months after hospital discharge followup visit (V2);
* the 6-to-12-months after hospital discharge followup visit, performed for study subjects that at V2 show clinical and/or functional and/or radiological abnormalities due to sequelae of COVID-19 (V3).

For data analysis, all variables will be analyzed using descriptive method. Continuous variables will be presented as means, standard deviation, median and respective minimum and maximum values; the discrete or nominal variables will be expressed as frequencies and relative percentages. Subgroup analysis will be performed using X- 2 test or Fischer test when appropriate; parametric variables not normally distributed will be analyzed by Kruskal-wallis non-parametric test. Association between two or more parameters will be calculate with Spearman Correlation. p <0.05 values will be considered statistically significant.

This study was approved by the Local Ethic Committee.

ELIGIBILITY:
Inclusion Criteria:

* acute respiratory failure due to SARS-COV-2 pneumonia
* sign of informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with SARS-COV-2 pneumonia discharged from our Insitution (Respiratory and Critical Care Unit - S.Orsola-Malpighi University Hospital, Bologna, IT) or patients referred to our Clinic for the followup of SARS-COV-2 pneumonia after hospital stay.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Long term evolution of clinical involvement due to SARS-COV-2 pneumonia / symptoms | from hospital stay to 6-to-12 months after hospital discharge for SARS-COV-2 pneumonia.
  For long term clinical evolution of SARS-COV-2 pneumonia Investigators will evaluate the presence or absence of each of the following symptoms (yes/no respectively for presence/absence):
  * dyspnea,
  * fatigue,
  * cough,
  * fever,
  * thoracic pain,
  * nausea,
  * diarrhea,
  * dysgeusia. The presence of each of these symptoms will be collected at the time of the hospital stay due to COVID-19 (H) and at 1-month after hospital discharge followup visit (V1); at 3-months after hospital discharge followup visit (V2); at 6-to-12-months after hospital discharge followup visit (V3). V3 will be performed for study subjects that at V2 show clinical and/or functional and/or radiological abnormalities due to sequelae of COVID-19.
  Differences in terms of presence and type of each symptoms between H, V1, V2 and V3 will be evaluated.
Long term evolution of clinical involvement due to SARS-COV-2 pneumonia / respiratory rate | from hospital stay to 6-to-12 months after hospital discharge for SARS-COV-2 pneumonia.
  For long term clinical evolution of SARS-COV-2 pneumonia Investigators will collect respiratory rate (RR, breaths/minute) of study subjects collected during the hospital stay due to COVID-19 (H); at V1, V2and V3. Difference in RR between H, V1, V2 and V3 will be evaluated.
Long term evolution of functional involvement due to SARS-COV-2 pneumonia - blood gas exchange parameters/partial pressure of oxygen and partial pressure of carbon monoxide | from hospital stay to 6-to-12 months after hospital discharge for SARS-COV-2 pneumonia
  Investigators will collect:
  * partial pressure of oxygen [paO2, mmHg],
  * partial pressure of carbon monoxide [paCO2 mmHg],
  emerged from blood gas exchange analysis performed during H, V1, V2 and V3. For each parameter (paO2, paCO2) the difference between value at H, V1,V2 and V3 will be evaluated.
Long term evolution of functional involvement due to SARS-COV-2 pneumonia - blood gas exchange parameters/ ph | from hospital stay to 6-to-12 months after hospital discharge for SARS-COV-2 pneumonia
  Investigators will collect:
  - ph [absolute value],
  emerged from blood gas exchange analysis performed during H, V1, V2 and V3. Difference between pH value at H, V1,V2 and V3 will be evaluated.
Long term evolution of functional involvement due to SARS-COV-2 pneumonia - blood gas exchange parameters/ oxygen saturation | from hospital stay to 6-to-12 months after hospital discharge for SARS-COV-2 pneumonia
  Investigators will collect:
  - oxygen saturation [SatO2, in %]),
  emerged from blood gas exchange analysis performed during H, V1, V2 and V3. Difference between SatO2 value at H, V1,V2 and V3 will be evaluated.
Long term evolution of functional involvement due to SARS-COV-2 pneumonia - blood gas exchange parameters: P/F ratio | from hospital stay to 6-to-12 months after hospital discharge for SARS-COV-2 pneumonia
  Investigators will collect:
  - P/F ratio (ratio between the measured paO2 and fraction of inspired oxygen ratio) expressed in absolute ratio;
  emerged from blood gas exchange analysis performed during H, V1, V2 and V3. Difference between P/F ratio value at H, V1,V2 and V3 will be evaluated.
Long term evolution of functional involvement due to SARS-COV-2 pneumonia - pulmonary function tests/ forced expiratory volume in the first second; forced vital capacity; total lung capacity; residual volume | from 1 month after hospital discharge for SARS-COV-2 pneumonia to 6-to-12 months after hospital discharge
  Investigators will consider the following parameters:
  * forced expiratory volume in the first second [FEV1,expressed in % of predicted value];
  * forced vital capacity [FVC, expressed in % of predicted value];
  * total lung capacity [TLC, expressed in % of predicted value];
  * residual volume [RV, expressed in % of predicted value];
  collected through pulmonary function tests performed at V1, V2 and V3. For each parameter (FEV1, FVC, TLC, RV) the difference between value at V1,V2 and V3 will be evaluated.
Long term evolution of functional involvement due to SARS-COV-2 pneumonia - pulmonary function tests/ FEV1/FVC ratio and RV/TLC ratio | from 1 month after hospital discharge for SARS-COV-2 pneumonia to 6-to-12 months after hospital discharge
  Investigators will consider the following parameters:
  * FEV1/FVC absolute ratio;
  * RV/TLC absolute ratio;
  collected through pulmonary function tests performed at V1, V2 and V3. For each parameter (FEV1/FVC, RV/TLC) the difference between value at V1,V2 and V3 will be evaluated.
Long term evolution of functional involvement due to SARS-COV-2 pneumonia - diffusing capacity of carbon monoxide | from 1 month after hospital discharge for SARS-COV-2 pneumonia to 6-to-12 months after hospital discharge
  Investigators will consider diffusing capacity of carbon monoxide (DLCO), expressed in % of the predicted value collected during V1, V2 and V3. Differences in terms of DLCO values between V1, V2 and V3 will be calculated.
Long term evolution of functional involvement due to SARS-COV-2 pneumonia - six minute walking test distance | from 1 month after hospital discharge for SARS-COV-2 pneumonia to 6-to-12 months after hospital discharge.
  Investigators will consider 6 minute walking test [6MWT] distance, expressed in meters collected during V1, V2 and V3. Differences in terms of 6MWT distance between V1, V2 and V3 will be calculated.
Long term evolution of functional involvement due to SARS-COV-2 pneumonia - presence of desaturation during six minute walking test | from 1 month after hospital discharge for SARS-COV-2 pneumonia to 6-to-12 months after hospital discharge.
  Investigators will consider the presence (yes/no) of desaturation at 6MWT (defined as a difference > 3% between baseline SatO2% and minimum SatO2% during test) collected during V1, V2 and V3. Differences in terms of presence of desaturation at 6MWT between V1, V2 and V3 will be calculated.
long term evolution of radiological involvement due to SARS-COV-2 pneumonia | from hospital stay to 6-to-12 months after hospital discharge for SARS-COV-2 pneumonia.
  For long term radiological evolution of SARS-COV-2 pneumonia Investigators will consider:
  * presence [yes/no] of consolidation and/or ground-glass opacities at chest X-ray and high resolution computed tomography (HRCT) of the lungs,
  * presence/absence [yes/no] of lung abnormalities in lung ultrasound (LUS) evaluation,
  collected each during H, V1, V2 and V3. Differences between H,V1,V2 and V3 for each characteristics will be described.

SECONDARY OUTCOMES:
identifying possible factors associated to the persistency of clinical, functional and radiological long term lung involvement due to COVID-19 | from hospital stay to 6-to-12 months after hospital discharge for SARS-COV-2 pneumonia.
  To identify possible factors associated or correlated to the persistency of clinical and/or functional and/or radiological long term lung involvement due to SARS-COV-2 pneumonia at V1, V2, V3, primary outcome measurements will be stratified according to:
  * the presence [yes/no] of comorbidities (cardiovascular, chronic obstructive pulmonary disease, asthma, immunological disorders, solid cancer, hematological malignancy, diabetes mellitus, immunodepression);
  * age (expressed in years, age≥60 versus age<60 years);
  * sex (male versus female);
  * hospital stay duration (expressed in days);
  * acute respiratory failure duration (expressed in days);
  of study subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory and Critical Care Unit - S.Orsola-Malpighi University Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No